CLINICAL TRIAL: NCT03296605
Title: Impacts of Bariatric Surgery on Obesity in China
Brief Title: Development of Obesity and Bariatric Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zhu DaLong, Director, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: AF/SC-08/02.0
Record Dates: First submitted 2017-09-12; First posted 2017-09-28 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Adipose tissue, Liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: Patients with obesity already received bariatric surgery
- Healthy control: Volunteers with normal body weight and already received abdominal surgery

SUMMARY:
This study focus on the cause of obesity and impacts of bariatric surgery on it.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index ≥18 kg/m2
2. already received bariatric surgery or abdonimal surgery

Exclusion Criteria:

1. acute stroke or acute myocardial infarction in 6 months
2. autoimmune disease
3. long-term use of non-steroidal anti-inflammatory drugs, corticosteroids and immunosuppressive drugs
4. pregnancy
5. consists with other endocrine diseases
6. acute infection in2 weeks
7. cancer
8. use of antibiotics in 3 months
9. chronic digestive inflammations 9

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obesity patients and controls
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Immunity cells | up to 5 years
  Ratio of immunity cells in circulating and adipose or liver tissue

SECONDARY OUTCOMES:
Body weight and height | up to 5 years
  Body weight and height will be combined to report BMI in kg/m^2
Insulin | up to 5 years
  Insulin (mIU/L) concentartions in serum and adipose tissue
Cytokine | up to 5 years
  Cytokines concentrations in circulating and adipose or liver tissue
Cognitive Assessment (MMSE) | up to five years
  Mini-Mental State Examination (MMSE) scores from 0-30, and the test means better cognition with a higher score.
Cognitive Assessment (MoCA) | up to 5 years
  The Montreal Cognitive Assessment (MoCA) scores from 0-30, and the test means better cognition with a higher score.
Cognitive Assessment (RBANS) | up to 5 years
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores from 0-800, and the test means better cognition with a higher score.
Cognitive Assessment (processing speed) | up to 5 years
  The Trial Making Test (TMT) provides a measure of processing speed, which consists of part A and part B (TMT-A and TMT-B). The time limits for performing the TMT-A and TMT-B are 180 and 300 seconds, respectively. Processing speed is estimated by the sum of the consuming time to complete TMT-A and TMT-B such that less time indicate faster processing speed.
Cognitive Assessment (executive function) | up to 5 years
  The Victoria Stroop Color-Word Test is a well-known measure of executive functioning. There are three indices including Stroop-dot, Stroop-word and Stroop-color word in the test. The color task consists of colored dots; the word task comprises ordinary words that are unrelated to the meaning of color; the color-word task consists of words written in color that indicate the meaning of the color, but the color of these words differs from the meaning of the word itself. The participants were asked to quickly read the color of the dots or Chinese words on the cards. The sum of consuming time taken to read the three cards is used as an index of executive function performance. Less time indicates better executive function.
brain structure and activation in fMRI | up to 5 years
  All patients underwent odor-induced task fMRI on a 3.0T MR scanner

CONTACTS AND LOCATIONS:
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Tang W, Ge K, Shen L, Wang H, Feng W, Sun X, Chu X, Zhu D, Yin H, Bi Y. Th1 bias of liver mucosal-associated invariant T cells promotes hepatic gluconeogenesis in type 2 diabetes mellitus. Diabetes Metab Res Rev. 2023 May;39(4):e3620. doi: 10.1002/dmrr.3620. Epub 2023 Feb 17. PMID 36738300
- [Derived] Liu F, He J, Liu B, Zhang P, Wang H, Sun X, Chu X, Guan W, Feng W, Bi Y, Zhu D. Association of Omental Adipocyte Hypertrophy and Fibrosis with Human Obesity and Type 2 Diabetes. Obesity (Silver Spring). 2021 Jun;29(6):976-984. doi: 10.1002/oby.23155. Epub 2021 May 4. PMID 33943025
- [Derived] Yuan X, Chen J, Cheng Q, Zhao Y, Zhang P, Shao X, Bi Y, Shi X, Ding Y, Sun X, Xue B. Hepatic expression of Yin Yang 1 (YY1) is associated with the non-alcoholic fatty liver disease (NAFLD) progression in patients undergoing bariatric surgery. BMC Gastroenterol. 2018 Oct 3;18(1):147. doi: 10.1186/s12876-018-0871-2. PMID 30285651
- [Derived] Zhang P, Ge Z, Wang H, Feng W, Sun X, Chu X, Jiang C, Wang Y, Zhu D, Bi Y. Prolactin improves hepatic steatosis via CD36 pathway. J Hepatol. 2018 Jun;68(6):1247-1255. doi: 10.1016/j.jhep.2018.01.035. Epub 2018 Feb 13. PMID 29452209